CLINICAL TRIAL: NCT00483158
Title: A Double-Blind, Placebo-Controlled, Randomized, Dose-Escalating Study of Single and Multiple Oral Doses of Finafloxacin Hydrochloride in Healthy Subjects and a Study of H. Pylori Treatment in Healthy Carriers
Brief Title: First Time in Man Study of Finafloxacin Hydrochloride
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MerLion Pharmaceuticals GmbH (Industry)
Responsible Party: Michael Seiberling, MD, Prinzipal Study Investigator, Swiss Pharma Contract, Basel, Switzerland
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FINA-001
Record Dates: First submitted 2007-06-04; First posted 2007-06-06 (Estimated); Last update posted 2008-07-29 (Estimated); Status verified 2008-07

CONDITIONS: Helicobacter Infections; Urinary Tract Infection
Keywords: Helicobacter pylori; Fluoroquinolones; First in Man
MeSH Terms: conditions — Helicobacter Infections; Urinary Tract Infections

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- A (Placebo Comparator): Rising Single Dose
  Interventions: Drug: Finafloxacin hydrochloride
- B (Placebo Comparator): Rising Multiple Dose
  Interventions: Drug: Finafloxacin hydrochloride
- C (Experimental): Open Label H. pylori cohort
  Interventions: Drug: Finafloxacin hydrochloride

INTERVENTIONS:
Drug: Finafloxacin hydrochloride — Tablets, oral single dose and multiple dose once daily for 7d

SUMMARY:
The purpose of this study is to study the safety of single doses and multiple doses of Finafloxacin hydrochloride in healthy volunteers. The level of Finafloxacin hydrochloride will be measured in the subjects blood and urine. One part of the study will assess if Finafloxacin hydrochloride eradicates Helicobacter pylori, a stomach bacteria. Another part of the study will assess the activity of the drug in urine.

DETAILED DESCRIPTION:
New antibiotics are needed due to the increasing resistance of bacteria to existing antibiotics. Helicobacter pylori (H. pylori) is a bacteria of the stomach and has been shown to cause peptic ulcers and is implicated in gastric cancer. Up to 40% of the population has H. pylori. Current treatments used to eradicate H. pylori are a combination of a number of drugs including antibiotics and drugs which reduce the acid in the stomach. These treatments are complicated and some H. pylori is resistant to the antibiotics used.

This study is the first use of Finafloxacin hydrochloride in man and will examine its safety and make a preliminary study of its effectiveness as a single agent in eradicating H. pylori. The urine of subjects will also be used to test its effectiveness in killing the bacteria which cause urinary tract infections.

ELIGIBILITY:
Inclusion Criteria:

* Male or female healthy subjects
* 18-55 years of age
* In good health
* For part C only, Helicobacter pylori carrier status as assessed by a positive result of the urease breath test at screening.

Exclusion Criteria:

* Abnormal physical findings of clinical significance at the Screening examination or baseline which would interfere with the objectives of the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 95 (Actual)
Dates: Start 2007-08; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of single and multiple oral doses of Finafloxacin HCl by assessing adverse events, physical examinations, clinical chemistry examination, hematology, ECG and urinalysis. | 7 days

SECONDARY OUTCOMES:
To determine the pharmacokinetic profile of single and multiple oral doses of Finafloxacin HCl in healthy subjects | 7 days
To determine the bactericidal activity of urine obtained from healthy subjects after administration of Finafloxacin HCl | 7 days
To explore the activity of multiple oral doses of Finafloxacin HCl against Helicobacter pylori using the effect on the urease breath test in healthy carriers as a model | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Michael Seiberling, MD, Principal Investigator — SWISS PHARMA CONTRACT LTD
Locations (1):
- Swiss Pharma Contract Ltd, Basel, Switzerland